CLINICAL TRIAL: NCT02572986
Title: A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% to Elimite™ Cream 5% in the Treatment of Scabies
Brief Title: A Study to Evaluate the Therapeutic Equivalence of Generic Permethrin Cream 5% to Elimite® in the Treatment of Scabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRL-USG02-P/2015
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Permethrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Permethrin cream 5% (Experimental): Manufactured by Dr. Reddy's Laboratories, Ltd
  Interventions: Drug: Permethrin
- Elimite™ Cream (permethrin) 5% (Active Comparator): Manufactured by Prestium Pharma, Inc
  Interventions: Drug: Permethrin

INTERVENTIONS:
Drug: Permethrin

SUMMARY:
Scabies is an infestation of the skin by the human itch mite (Sarcoptes scabiei). Diagnosis of scabies is made based on clinical symptoms, such as nocturnal itching, and appearance and distribution of the rash. Definitive diagnosis includes the microscopic identification of the mite, mite eggs, or mite fecal matter in the skin. Topical permethrin is considered the drug of choice for the treatment of scabies. It is a synthetic pyrethroid that is safe for use in adults and children 2 months and older.

This study will evaluate the therapeutic equivalence of a generic permethrin cream 5% to Elimite® in the Treatment of Scabies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent that meets all criteria of current FDA regulations.
2. Male or non-pregnant, non-lactating female at least 2 years of age or older.
3. Diagnosis of active scabies by presence of a burrow and/or typical scabietic lesions at the classic sites of infestation.
4. Parasitological confirmation of clinical diagnosis with demonstration under light microscope of mites and/or their products (larvae, eggs or fecal material).
5. Symptom score of 2 or 3 on a 4-point rating scale of 0-3 for nocturnal itching.
6. Women must be either 1 year post-menopausal (no menstrual periods for at least 12 months), surgically sterile, or if they are of child-bearing potential, they must:

   * Have been using systemic birth control, intrauterine device, or used barrier methods such as diaphragm plus spermicide or condom plus spermicide consistently, at least 14 days before study cream administration.
   * Had a normal menstrual cycle for the month before start of treatment.
   * Have a negative urine pregnancy test result upon entry into the study.
   * Agree to use a medically accepted form of birth control (oral, implant, injectable or transdermal contraceptives, intrauterine device, condom plus spermicide, diaphragm plus spermicide) or practice abstinence throughout the study period.
7. Free from any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events.
8. Ability to apply study product to self or to other person if a child. If patient is a child, then parent/guardian will apply study product to him/her.

Exclusion Criteria:

1. Known hypersensitivity to permethrin cream or any of its components, ragweed or chrysanthemums, synthetic pyrethroids or pyrethrin.
2. Use of any systemic or topical acaricide 1 month before enrollment.
3. Patients with crusted/Norwegian scabies.
4. Patients with an underlying immunodeficient state (including prolonged treatment with corticosteroids), immunosuppressive disorders requiring therapy, severe systemic disease and history of HIV infection.
5. Any condition, medical, psychological, or social, that, in the Investigator's opinion, would interfere with participation in the study.
6. Women who are pregnant, planning pregnancy or lactating.
7. Family members of employees of the clinic or Investigator.
8. Patients who, in the opinion of the Investigator, would be non-compliant with the requirements of the study protocol.
9. Patients whose close personal contacts will not or are not willing to comply with standard of care for Scabies management.
10. Patients less than 2 years of age.
11. Patients or guardians of patients, who are unable or unwilling to give informed consent or assent respectively.
12. Receipt of any drug as part of a research study within 30 days before screening.
13. History of seizures.
14. Severe cutaneous bacterial or fungal infections requiring therapy (including systemic and topical antibiotics) or coexisting dermatological disorder that could interfere with the diagnosis and subsequent monitoring of scabies.
15. Treatment with systemic or topical corticosteroids less than 2 weeks and less than 1 week from enrollment, respectively.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with therapeutic cure (parasitological cure plus clinical cure) of scabies | Day 28

SECONDARY OUTCOMES:
The proportion of patients with no itch persistence | Day 28

OTHER OUTCOMES:
Adverse events assessment | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ashis Patnaik, MD, Study Director — Dr. Reddy's Laboratories Limited; Prasanna Ganapathi, MD, Study Director — Dr. Reddy's Laboratories Limited; Shilpi Dhawan, MD, Study Director — Dr. Reddy's Laboratories Limited
Locations (13):
- United States (10):
  - Omni Dermatology, Phoenix, Arizona
  - Sun Rise Clinical Research, Inc, Bell Gardens, California
  - Havana Research Institute, Pasadena, California
  - Solutions Through Advanced Research, Jacksonville, Florida
  - San Marcus Research Clinic, Incorporation, Miami, Florida
  - L & C Professional Medical Research Institute, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Derm Dx Center for Dermatology, Hazleton, Pennsylvania
  - Sun Research Institute, San Antonio, Texas
  - Zain Research, LLC, Richland, Washington
- El Salvador (2):
  - Clinica Dermatologica, San Salvador
  - Clinica Dermatologica y Cirugia de Piel, Santa Tecla, La Libertad
- Clinica Dermatologica Dra. Yariela Grajales, Panama City, PanamaCity, Panama